CLINICAL TRIAL: NCT04647786
Title: Safe and Effective Above Cuff Tracheostomy Ventilation - a Device Development Study
Brief Title: Safe and Effective Above Cuff Tracheostomy Ventilation
Acronym: SEACtV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Manchester Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: B00990
Record Dates: First submitted 2020-11-20; First posted 2020-12-01 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Tracheostomy

STUDY DESIGN:
Intervention Model Description: 3 phases:
  1. Safety testing in sequential patients
  2. 2x2 factorial design
  3. Simple unblinded RCT using finalised device vs standard care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Humidified and Augmented gas flows (Experimental)
  Interventions: Device: Prototype medical device (SEA CtV)
- Humidified but not Augmented gas flows (Experimental)
  Interventions: Device: Prototype medical device (SEA CtV)
- Not Humidified but Augmented gas flows (Experimental)
  Interventions: Device: Prototype medical device (SEA CtV)
- Neither humidified nor augmented gas flows (No Intervention)
- Use of finalised device (SEA CtV) in final phase (Experimental)
  Interventions: Device: Prototype medical device (SEA CtV)
- Standard care (no SEA CtV) (No Intervention)

INTERVENTIONS:
Device: Prototype medical device (SEA CtV) — A prototype device that delivers a controlled flow of gas to the upper airways via the subglottic suction port of an established tracheostomy tube. Gas flow may be timed, warmed and/or humidified.
  Arms: Humidified and Augmented gas flows; Humidified but not Augmented gas flows; Not Humidified but Augmented gas flows; Use of finalised device (SEA CtV) in final phase

SUMMARY:
A Phase I study of an 'in-house' developed, novel, Class I, prototype medical device to facilitate vocalisation in participants with cuff-inflated tracheostomy tubes.

Primary objective: To design and develop a device to deliver Above Cuff Vocalisation (ACV) that is safe, well tolerated and effective at producing a voice in tracheostomised patients in the Intensive Care Unit (ICU).

Secondary objective: To evaluate whether more effective delivery of ACV has a significant impact on laryngeal function and recovery following new tracheostomy in ICU patients.

DETAILED DESCRIPTION:
A tracheostomy is an artificial airway inserted into the trachea (windpipe) through the front of the neck, usually required for prolonged artificial ventilation in the critically ill. Between 10-15% of the 250,000 patients admitted annually to UK Intensive Care Units (ICUs) require temporary tracheostomy, with an additional 5,000 tracheostomies performed during surgery. The tubes have a cuff/balloon which seals the trachea when inflated, allowing lung ventilation. The flow of gas into and out of the patient's lungs does not flow through the upper airways (nose and mouth), bypassing the larynx (voice box) and preventing speech. Our research found the biggest problem with tracheostomies from the patient's perspective is losing the ability to speak. If the muscles of the larynx and throat are not used, they quickly become weak, meaning that coughing, swallowing and talking can take longer to recover. These problems cause anger, frustration, fear and low mood and lead to significantly longer hospital stays, impacting ICU and hospital bed availability.

Patients with a weak cough or swallow cannot clear secretions from the throat, which may enter the lungs (aspiration). The inflated cuff reduces aspiration and most ICU-specific tubes have an extra suction-port for secretion removal. However, additional gas can be directed via the suction-port, through the vocal cords and out via the upper airways, allowing vocalisation. The MHRA confirmed these tubes can be used for 'above cuff voicing' (ACV) in line with their CE marking.

Our proposed research advances healthcare technologies by developing a new clinically validated prototype medical device with the potential to significantly increase patient benefit for a defined and expanding area of clinical need. Our collaborative project combines our clinical experience and understanding of the needs of tracheostomy patients and their families with the design and engineering excellence of our University and SME partners. Our team is supported by individual and institutional research expertise and together with our patient partners, we can deliver an advanced prototype device with a clear pathway towards adoption and commercialisation, attractive to follow-on funders and investors.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria (patient):

* Provision of informed consent prior to any study specific procedures
* cuff-inflated tracheosotmy tube in situ for >48 hours
* managed on an Intensive Care Unit at MFT
* Male and females
* Aged 18-100; patient is alert and attempting to communicate (and thus able to participate in the consent process).

Inclusion criteria (staff):

* Provision of informed consent
* bedside clinical staff (medical, nursing, allied healthcare professional) who manage the patient during routine clinical duties whilst ACV is in progress.

Exclusion Criteria:

Exclusion criteria (patient): Participants must not enter the study if any of the following exclusion criteria are fulfilled:

* Patient refusal
* ACV is not indicated in the opinion of the parent clinical team
* Patient has (or is suspected to have) an altered and therefore potentially obstructed upper airway
* Patient has (or is suspected to have) an active and currently infectious high-consequence respiratory infection that could be transmitted by aerosolisation (eg COVID-19)
* Clinical condition has progressed so that the patient is tolerating cuff deflation and a speaking valve well and is able to voice effectively (ie without ACV: this negates the requirement for an ACV trial); Contraindications to FEES (adapted from RCSLT FEES policy) o Base of skull / facial fracture; Severe/life threatening epistaxis within the last 6 weeks; Trauma to nasal cavity secondary to surgery or injury within the last 6 weeks; Sino-nasal and anterior skull base tumours / surgery; Nasopharyngeal stenosis; Craniofacial anomalies; Hereditary Haemorrhagic telangiectasia

Exclusion criteria (staff): Refusal to participate.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness of vocalisation (Patient-reported voice VAS) | Daily for up to 7 days
  To assess the effectiveness of the SEA CtV prototype device in producing a voice for cuff-inflated tracheostomy patients.

SECONDARY OUTCOMES:
Voice rating | Daily for up to 7 days
  (Objective scales FCS, NoWS, TOMS, GRBAS, recordings for volume and intelligibility); Cough count; Swallow count; e-Stim (threshold/max sensetivities); FEES (Laryngeal function scales Pen-Asp, SSRS, APS)
Adverse events record | Daily for up to 7 days
  Adverse events record (tracheosotmy tube displacement, surgical emphysema), adverse events log, setup safety tests (does the device stop appropriately)
Patient reported subjective tolerability | Daily for up to 7 days
  Patient-reported subjective tolerability VAS; Staff-reported objective tolerability VAS; Patient-reported problems; ACV device use
Time to first oral intake | Daily for up to 7 days
  Time to oral intake; Functional Swallowing Outcome; vocalisation; cuff deflation for >2 hours; ETT days; Trachy days; ICU days; hospital days; CCMDS organ supoort data

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The project will generate confidential patient data and commercially sensitive IP data. Summaries of these data will be shared publicly.

REFERENCES:
- [Background] McGrath BA, Wallace S, Wilson M, Nicholson L, Felton T, Bowyer C, Bentley AM. Safety and feasibility of above cuff vocalisation for ventilator-dependant patients with tracheostomies. J Intensive Care Soc. 2019 Feb;20(1):59-65. doi: 10.1177/1751143718767055. Epub 2018 Mar 28. PMID 30792764
- [Background] Zaga CJ, Pandian V, Brodsky MB, Wallace S, Cameron TS, Chao C, Orloff LA, Atkins NE, McGrath BA, Lazarus CL, Vogel AP, Brenner MJ. Speech-Language Pathology Guidance for Tracheostomy During the COVID-19 Pandemic: An International Multidisciplinary Perspective. Am J Speech Lang Pathol. 2020 Aug 4;29(3):1320-1334. doi: 10.1044/2020_AJSLP-20-00089. Epub 2020 Jun 11. PMID 32525695
- [Background] McGrath B, Lynch J, Wilson M, Nicholson L, Wallace S. Above cuff vocalisation: A novel technique for communication in the ventilator-dependent tracheostomy patient. J Intensive Care Soc. 2016 Feb;17(1):19-26. doi: 10.1177/1751143715607549. Epub 2015 Oct 5. PMID 28979454
- See also: UK National Tracheostomy Safety Project webpage and video demonstrating the problem and current solution — http://www.tracheostomy.org.uk/healthcare-staff/vocalisation/acv-above-cuff-vocalisation